CLINICAL TRIAL: NCT04644328
Title: The Doctors for Coronavirus Prevention Project Thanksgiving / Christmas Messaging Campaign
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Bureau of Economic Research, Inc. (Other)
Collaborators: Massachusetts Institute of Technology (Other); Harvard University (Other); Massachusetts General Hospital (Other); Yale University (Other); Stanford University (Other)
Responsible Party: Principal Investigator, Esther Duflo, Abdul Latif Jameel Professor of Poverty Alleviation and Development Economics, MIT; Co-Director, Abdul Latif Jameel Poverty Action Lab, National Bureau of Economic Research, Inc.
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 2003000118A010
Record Dates: First submitted 2020-11-13; First posted 2020-11-25 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: A total of 13 states, comprising 829 counties, centrally report COVID-19 cases at the ZCTA level. Two separate experiments were run within the study, one around Thanksgiving and one around Christmas. For each experiment, approximately half of the counties were randomized to high-intensity treatment with the remaining randomized to low-intensity treatment. In high-intensity counties, 3/4 of ZCTAs were treated and 1/4 were not. In low-intensity counties, 1/4 of ZCTAs were treated and 3/4 were not. In treated ZCTAs, Facebook users received ads with messages from physicians and other health personnel urging them to stay home and wear masks to stop the spread of COVID-19. Users in non-treated ZCTAs received no such ads. After exclusions, 820 counties were randomized to high- or low-intensity treatment during Thanksgiving and 767 counties were during Christmas.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Intensity Treatment Arm (Experimental): Treatment: Individuals received approximately 3 Facebook ads over a 2-week period. Each ad contained a short video recorded by a physician using a script that discusses staying safe during the holidays by considering not traveling and using a mask when appropriate.
  Randomization to treatment: The 13 states which centrally report COVID-19 cases at the ZCTA level contained 829 counties. At Thanksgiving, 9 counties were excluded due to data limitations. At Christmas, 62 counties were excluded due to data limitations and potential negative impacts in rural, conservative areas resulting from polarization in the wake of the 2020 presidential election. Approximately half of the counties were randomized to high-intensity treatment with the remaining randomized to low-intensity treatment. In high-intensity counties, 3/4 of ZCTAs were treated (i.e., Facebook users in those ZCTAs received ads) and 1/4 were not. In low-intensity counties, 1/4 of ZCTAs were treated and 3/4 were not.
  Interventions: Behavioral: Facebook Ads on the importance of staying safe during the Thanksgiving / Christmas holiday
- Low-Intensity Control Arm (No Intervention): Control: Individuals did not receive ads containing short physician-recorded videos.
  Randomization to treatment: The 13 states which centrally report COVID-19 cases at the ZCTA level contained 829 counties. At Thanksgiving, 9 counties were excluded due to data limitations. At Christmas, 62 counties were excluded due to data limitations and potential negative impacts in rural, conservative areas resulting from polarization in the wake of the 2020 presidential election. Approximately half of the counties were randomized to high-intensity treatment with the remaining randomized to low-intensity treatment. In high-intensity counties, 3/4 of ZCTAs were treated (i.e., Facebook users in those ZCTAs received ads) and 1/4 were not. In low-intensity counties, 1/4 of ZCTAs were treated and 3/4 were not.

INTERVENTIONS:
Behavioral: Facebook Ads on the importance of staying safe during the Thanksgiving / Christmas holiday — Facebook ads to show a 15 second video clip recorded by MGH, Harvard and Lynn Community health center and other health care professionals. The ads will be shown before the Thanksgiving/Christmas holiday and will focus on staying safe - limiting travel and mask-wearing. The investigators will randomize exposure to the ad campaign at the ZIP code or county level.
  Arms: High-Intensity Treatment Arm

SUMMARY:
Facebook ads with physician-delivered videos were shown before the Thanksgiving and Christmas holidays and focused on staying safe during the COVID pandemic by limiting travel and mask-wearing.

DETAILED DESCRIPTION:
The investigators used Facebook ads to show a 20 second video clip recorded by Massachusetts General Hospital, Harvard and Lynn Community health center doctors (6 people in all) to approximately 20,000,000 Facebook users. The ads will be shown before the Thanksgiving and Christmas holiday and will focus on staying safe - limiting travel and mask-wearing. The investigators will randomize exposure to the ad campaign at the ZIP code or county level to ask:

Do the videos change mobility and Thanksgiving and Christmas holiday travel? Do they reduce the spread of COVID-19?

Are there spillover impacts from the video messages? For example, if individuals decide to stay home, then do the geographical regions that tend to be visited by people from treated areas experience any effects, either through information spillovers or through a reduction in travel?

ELIGIBILITY:
Inclusion Criteria:

- Individuals viewing the ads must be Facebook users, 18 years and older. Facebook will decide specifically which users receive the messages within a target geographical area (zip or county).

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 820 (Actual)
Dates: Start 2020-11-12 (Actual); Primary Completion 2021-02-11 (Actual); Study Completion 2021-02-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- JPAL North America, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
The pre-analysis plan will be posted publicly. The ability to share IPD will be based on discussions with our partner organization.

REFERENCES:
- [Result] Breza E, Stanford FC, Alsan M, Alsan B, Banerjee A, Chandrasekhar AG, Eichmeyer S, Glushko T, Goldsmith-Pinkham P, Holland K, Hoppe E, Karnani M, Liegl S, Loisel T, Ogbu-Nwobodo L, Olken BA, Torres C, Vautrey PL, Warner ET, Wootton S, Duflo E. Effects of a large-scale social media advertising campaign on holiday travel and COVID-19 infections: a cluster randomized controlled trial. Nat Med. 2021 Sep;27(9):1622-1628. doi: 10.1038/s41591-021-01487-3. Epub 2021 Aug 19. PMID 34413518

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The 13 states which centrally report COVID-19 cases at the ZCTA level contained 829 counties. At Thanksgiving, 9 counties were excluded due to data limitations; at Christmas, 62 counties were excluded due to data limitations and potential negative impacts of treatment in rural, conservative areas resulting from polarization in the wake of the 2020 presidential election.
Units Other Than Participants: Counties
Groups:
- High-Intensity Counties: Treatment: Individuals received approximately 3 Facebook ads over a 2-week period. Each ad contained a short video recorded by a physician using a script that discusses the importance of staying safe during Thanksgiving or Christmas by considering not traveling and using a mask when appropriate.
  Randomization to treatment: The investigators randomized exposure to the ad campaign as follows. The 13 states which centrally report COVID-19 cases at the ZCTA level contained 829 counties. At Thanksgiving, 9 counties were excluded due to data limitations; at Christmas, 62 counties were excluded due to data limitations and potential negative impacts of treatment in rural, conservative areas resulting from polarization in the wake of the 2020 presidential election. Approximately half of the counties were randomized to high-intensity treatment with the remaining randomized to low-intensity treatment. In high-intensity counties, 3/4 of ZCTAs were treated (i.e., Facebook users in those ZCTAs received ads) and 1/4 were not. In low-intensity counties, 1/4 of ZCTAs were treated and 3/4 were not.
- Low-Intensity Counties: Control: Individuals did not receive ads containing short physician-recorded videos.
  Randomization to treatment: The investigators randomized exposure to the ad campaign as follows. The 13 states which centrally report COVID-19 cases at the ZCTA level contained 829 counties. At Thanksgiving, 9 counties were excluded due to data limitations; at Christmas, 62 counties were excluded due to data limitations and potential negative impacts of treatment in rural, conservative areas resulting from polarization in the wake of the 2020 presidential election. Approximately half of the counties were randomized to high-intensity treatment with the remaining randomized to low-intensity treatment. In high-intensity counties, 3/4 of ZCTAs were treated (i.e., Facebook users in those ZCTAs received ads) and 1/4 were not. In low-intensity counties, 1/4 of ZCTAs were treated and 3/4 were not.
Period: Thanksgiving Period
Arm/Group | High-Intensity Counties | Low-Intensity Counties
Started | NA; 410 Counties (Two separate, sequential experiments were run within the study using the same counties (with differences in exclusion criteria explained in the pre-assignment details). Thanksgiving experiment: 410 counties were assigned to high-intensity treatment. A total of 3,545 ZCTAs (of which 2,702 were in high-intensity counties) were treated. Counties randomized to intervention, data collected at the population level, actual number of participants unknown.) | NA; 410 Counties (Two separate, sequential experiments were run within the study using the same counties (with differences in exclusion criteria explained in the pre-assignment details). Thanksgiving experiment: 410 counties were assigned to low-intensity treatment. A total of 3,453 ZCTAs (of which 2,549 were in low-intensity counties) were not treated. Counties randomized to intervention, data collected at the population level, actual number of participants unknown.)
Completed | NA; 410 Counties (Counties randomized to intervention, data collected at the population level, actual number of participants unknown.) | NA; 410 Counties (Counties randomized to intervention, data collected at the population level, actual number of participants unknown.)
Not Completed | NA; 0 Counties | NA; 0 Counties
Period: Christmas Period
Arm/Group | High-Intensity Counties | Low-Intensity Counties
Started | NA; 386 Counties (Two separate, sequential experiments were run within the study using the same counties (with differences in exclusion criteria explained in the pre-assignment details). Christmas experiment: 386 counties were assigned to high-intensity treatment. A total of 5,077 ZCTAs (of which 3,818 were in high-intensity counties) were treated. Counties randomized to intervention, data collected at the population level, actual number of participants unknown.) | NA; 381 Counties (Two separate, sequential experiments were run within the study using the same counties (with differences in exclusion criteria explained in the pre-assignment details). Christmas experiment: 381 counties were assigned to low-intensity treatment. A total of 5,102 ZCTAs (of which 3,833 were in low-intensity counties) were not treated. Counties randomized to intervention, data collected at the population level, actual number of participants unknown.)
Completed | NA; 386 Counties (Counties randomized to intervention, data collected at the population level, actual number of participants unknown.) | NA; 381 Counties (Counties randomized to intervention, data collected at the population level, actual number of participants unknown.)
Not Completed | NA; 0 Counties | NA; 0 Counties

BASELINE CHARACTERISTICS:
Population: The experiment was run during two periods: Thanksgiving (Period 1) and Christmas (Period 2). During Thanksgiving, 820 counties were analyzed (410 high-intensity, 410 low-intensity). Of these counties, 767 were analyzed during Christmas (386 high-intensity, 381 low-intensity). Fewer counties were analyzed at Christmas because we removed counties in rural, conservative areas from the study due to potential negative impacts resulting from polarization in the wake of the 2020 presidential election.
Units Other Than Participants: Counties
Groups:
- Total: Total of all reporting groups
Arm/Group | High-Intensity Counties | Low-Intensity Counties | Total
Number analyzed (Participants) | NA | NA | NA
Number analyzed (Counties) | 410 | 410 | 820
Age, Customized [Mean (Standard Deviation); unit: Counties] — Population: Age data were not collected because no participants were enrolled.
  Counties
    number analyzed (Counties) | 0 | 0 | 0
Sex/Gender, Customized [Mean (Standard Deviation); unit: Counties] — Population: Sex/gender data were not collected because no participants were enrolled.
  Counties
    number analyzed (Counties) | 0 | 0 | 0
Race/Ethnicity, Customized [Mean (Standard Deviation); unit: Proportion] — Population: Race/ethnicity data were not collected because no participants were enrolled.
  Proportion
    Thanksgiving (Period 1) | NA (NA) — Race/ethnicity data were not collected because no participants were enrolled. | NA (NA) — Race/ethnicity data were not collected because no participants were enrolled. | NA (NA) — Race/ethnicity data were not collected because no participants were enrolled.
    Christmas (Period 2): number analyzed (Counties) | 386 | 381 | 767
    Christmas (Period 2) | NA (NA) — Race/ethnicity data were not collected because no participants were enrolled. | NA (NA) — Race/ethnicity data were not collected because no participants were enrolled. | NA (NA) — Race/ethnicity data were not collected because no participants were enrolled.
Baseline movement metric [Mean (Standard Deviation); unit: Percent change relative to Feb 2020] — Percent change in distance traveled by Facebook users in the county from Feb-Nov 2020 Population: Fewer counties were analyzed at Christmas because counties in rural, conservative areas from the study were removed from the study due to potential negative impacts resulting from polarization in the wake of the 2020 presidential election.
  Percent change relative to Feb 2020
    Thanksgiving (Period 1) | -8.58 (7.10) | -8.88 (6.42) | -8.73 (6.77)
    Christmas (Period 2): number analyzed (Counties) | 386 | 381 | 767
    Christmas (Period 2) | -8.69 (6.88) | -9.09 (6.56) | -8.89 (6.72)
Baseline leave home [Mean (Standard Deviation); unit: Percentage] — Percentage of Facebook users in a given county leaving their homes on Nov 13 2020 Population: Fewer counties were analyzed at Christmas because counties in rural, conservative areas from the study were removed from the study due to potential negative impacts resulting from polarization in the wake of the 2020 presidential election.
  Percentage
    Thanksgiving (Period 1) | 82.33 (2.42) | 82.49 (2.53) | 82.41 (2.47)
    Christmas (Period 2): number analyzed (Counties) | 386 | 381 | 767
    Christmas (Period 2) | 82.40 (2.43) | 82.44 (2.40) | 82.42 (2.41)
Missing baseline Facebook outcomes [Mean (Standard Deviation); unit: Proportion of counties] — Proportion of counties with missing Facebook baseline mobility data. To protect user privacy, Facebook does not release data in counties with a low number of users so not all counties will have baseline mobility data. Population: Fewer counties were analyzed at Christmas because counties in rural, conservative areas from the study were removed from the study due to potential negative impacts resulting from polarization in the wake of the 2020 presidential election.
  Proportion of counties
    Thanksgiving (Period 1) | 0.13 (0.34) | 0.17 (0.38) | 0.15 (0.36)
    Christmas (Period 2): number analyzed (Counties) | 386 | 381 | 767
    Christmas (Period 2) | 0.11 (0.32) | 0.13 (0.33) | 0.12 (0.32)
Baseline fortnightly cases [Mean (Standard Deviation); unit: Individuals] — Number of COVID-19 cases in the fortnight prior to baseline date Population: Fewer counties were analyzed at Christmas because counties in rural, conservative areas from the study were removed from the study due to potential negative impacts resulting from polarization in the wake of the 2020 presidential election.
  Individuals
    Thanksgiving (Period 1) | 683.90 (3,032.94) | 496.70 (1,165.17) | 590.30 (2,297.94)
    Christmas (Period 2): number analyzed (Counties) | 386 | 381 | 767
    Christmas (Period 2) | 654.77 (3,067.53) | 598.54 (1,343.02) | 626.84 (2,371.71)
Baseline fortnightly deaths [Mean (Standard Deviation); unit: Individuals] — Number of COVID-19 deaths in the fortnight prior to baseline date Population: Fewer counties were analyzed at Christmas because counties in rural, conservative areas from the study were removed from the study due to potential negative impacts resulting from polarization in the wake of the 2020 presidential election.
  Individuals
    Thanksgiving (Period 1) | 5.51 (22.35) | 4.64 (11.08) | 5.07 (17.63)
    Christmas (Period 2): number analyzed (Counties) | 386 | 381 | 767
    Christmas (Period 2) | 5.70 (23.07) | 5.07 (11.29) | 5.38 (18.19)
Share urban [Mean (Standard Deviation); unit: Proportion of county ZCTAs] — Proportion of zip code tabulation areas (ZCTAs) in county classified as urban. Urbanicity is defined per classifications released by the Federal Statistical System of the United States. Population: Fewer counties were analyzed at Christmas because counties in rural, conservative areas from the study were removed from the study due to potential negative impacts resulting from polarization in the wake of the 2020 presidential election.
  Proportion of county ZCTAs
    Thanksgiving (Period 1) | 0.47 (0.34) | 0.44 (0.34) | 0.46 (0.34)
    Christmas (Period 2): number analyzed (Counties) | 386 | 381 | 767
    Christmas (Period 2) | 0.48 (0.33) | 0.50 (0.33) | 0.49 (0.33)
Share Democrats [Mean (Standard Deviation); unit: Proportion of county voters] — Proportion of county voters who voted for the Democratic presidential candidate in 2020 Population: Fewer counties were analyzed at Christmas because counties in rural, conservative areas from the study were removed from the study due to potential negative impacts resulting from polarization in the wake of the 2020 presidential election.
  Proportion of county voters
    Thanksgiving (Period 1) | 0.36 (0.15) | 0.35 (0.15) | 0.36 (0.15)
    Christmas (Period 2): number analyzed (Counties) | 386 | 381 | 767
    Christmas (Period 2) | 0.37 (0.15) | 0.37 (0.15) | 0.37 (0.15)
Share Republicans [Mean (Standard Deviation); unit: Proportion of county voters] — Proportion of county voters who voted for the Republican presidential candidate in 2020 Population: Fewer counties were analyzed at Christmas because counties in rural, conservative areas from the study were removed from the study due to potential negative impacts resulting from polarization in the wake of the 2020 presidential election.
  Proportion of county voters
    Thanksgiving (Period 1) | 0.62 (0.16) | 0.63 (0.15) | 0.62 (0.15)
    Christmas (Period 2): number analyzed (Counties) | 386 | 381 | 767
    Christmas (Period 2) | 0.61 (0.15) | 0.61 (0.15) | 0.61 (0.15)
Population in 2019 [Mean (Standard Deviation); unit: individuals] — Population: Fewer counties were analyzed at Christmas because counties in rural, conservative areas from the study were removed from the study due to potential negative impacts resulting from polarization in the wake of the 2020 presidential election.
  individuals
    Thanksgiving (Period 1) | 122,491 (349,501) | 102,818 (282,369) | 112,654 (317,672)
    Christmas (Period 2): number analyzed (Counties) | 386 | 381 | 767
    Christmas (Period 2) | 116,787 (344,511) | 122,875 (309,239) | 119,811 (327,266)

OUTCOME MEASURES:

1. Primary Outcome: Facebook Movement Metric
Description: The change in movement metric is the percent change in distance covered in a day compared to the same day of the week in the benchmark period of February 2-29, 2020, by people who started the day in a particular location. We define holiday travel as travel during the three days preceding each holiday, since the available data does not allow us to compute the impact of the intervention on the return travel (after the holiday). The reason is that the mobility data describes the behavior throughout the day, for people who were in each county that morning. Since the campaign was targeted based on home location, we can only capture its impact on travel away from home, not back home.
Time Frame: November 26, 2020 (Thanksgiving); December 24-25, 2020 (Christmas); February 2-29, 2020 (Baseline benchmark)
Population: Rural, conservative counties were excluded during Christmas due to potential negative impacts of treatment resulting from polarization in the wake of the 2020 presidential election. The two periods have been entered as rows to avoid double-counting counties.
Measure: Mean (95% Confidence Interval); unit: Percent change relative to Feb 2020
Units Other Than Participants: Counties
Arm/Group | High-Intensity Counties | Low-Intensity Counties
Number analyzed (Participants) | NA | NA
Number analyzed (Counties) | 356 | 340
Percent change relative to Feb 2020
  Thanksgiving (Period 1) | -6.082 [-6.822 to -5.341] | -5.320 [-6.113 to -4.527]
  Christmas (Period 2): number analyzed (Counties) | 343 | 333
  Christmas (Period 2) | -2.603 [-3.279 to -1.927] | -1.823 [-2.588 to -1.057]

2. Primary Outcome: Percentage Leaving Home on Day of Holiday
Description: The Facebook stay put metric is the percentage of people who stay within a small geographical area (a "tile" of 600m*600m in which they started the day). We use it to compute the share of people leaving home on the day of the holiday (i.e. this variable = 1 - stay put on the day of the holiday).
Time Frame: November 26, 2020 (Thanksgiving); December 24-25, 2020 (Christmas)
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: Percentage
Units Other Than Participants: Counties
Arm/Group | High-Intensity Counties | Low-Intensity Counties
Number analyzed (Participants) | NA | NA
Number analyzed (Counties) | 356 | 340
Percentage
  Thanksgiving (Period 1) | 71.308 [70.885 to 71.731] | 71.468 [71.071 to 71.866]
  Christmas (Period 2): number analyzed (Counties) | 343 | 333
  Christmas (Period 2) | 72.859 [72.507 to 73.210] | 72.852 [72.520 to 73.185]

3. Primary Outcome: Inverse Hyperbolic Sine of COVID-19 Cases
Description: Inverse hyperbolic sine of COVID-19 cases during a 14 day period starting 5 days after each holiday
Time Frame: December 1-14 (Thanksgiving arms) and January 1-14 (Christmas arms)
Population: ZCTAs in rural, conservative counties were excluded during Christmas due to potential negative impacts of treatment resulting from polarization in the wake of the 2020 presidential election. The two periods have been entered as rows to avoid double-counting ZCTAs. Note that there are more ZCTAs in the Christmas control than Thanksgiving control because the two periods were randomized separately and the number of ZCTAs varies by county.
Measure: Mean (95% Confidence Interval); unit: Inverse hyperbolic sine of individuals
Units Other Than Participants: ZCTA
Groups:
- Treatment ZCTAs: Treatment: Individuals received approximately 3 Facebook ads over a 2-week period. Each ad contained a short video recorded by a physician using a script that discusses the importance of staying safe during Thanksgiving or Christmas by considering not traveling and using a mask when appropriate.
  Randomization to treatment: The investigators randomized exposure to the ad campaign as follows. The 13 states which centrally report COVID-19 cases at the ZCTA level contained 829 counties. At Thanksgiving, 9 counties were excluded due to data limitations; at Christmas, 62 counties were excluded due to data limitations and potential negative impacts of treatment in rural, conservative areas resulting from polarization in the wake of the 2020 presidential election. Approximately half of the counties were randomized to high-intensity treatment with the remaining randomized to low-intensity treatment. In high-intensity counties, 3/4 of ZCTAs were treated (i.e., Facebook users in those ZCTAs received ads) and 1/4 were not. In low-intensity counties, 1/4 of ZCTAs were treated and 3/4 were not.
- Control ZCTAs: Control: Individuals did not receive ads containing short physician-recorded videos.
  Randomization to treatment: The investigators randomized exposure to the ad campaign as follows. The 13 states which centrally report COVID-19 cases at the ZCTA level contained 829 counties. At Thanksgiving, 9 counties were excluded due to data limitations; at Christmas, 62 counties were excluded due to data limitations and potential negative impacts of treatment in rural, conservative areas resulting from polarization in the wake of the 2020 presidential election. Approximately half of the counties were randomized to high-intensity treatment with the remaining randomized to low-intensity treatment. In high-intensity counties, 3/4 of ZCTAs were treated (i.e., Facebook users in those ZCTAs received ads) and 1/4 were not. In low-intensity counties, 1/4 of ZCTAs were treated and 3/4 were not.
Arm/Group | Treatment ZCTAs | Control ZCTAs
Number analyzed (Participants) | NA | NA
Number analyzed (ZCTA) | 3427 | 3387
Inverse hyperbolic sine of individuals
  Thanksgiving (Period 1): number analyzed (ZCTA) | 3427 | 3346
  Thanksgiving (Period 1) | 4.333 [4.278 to 4.388] | 4.298 [4.243 to 4.353]
  Christmas (Period 2): number analyzed (ZCTA) | 3329 | 3387
  Christmas (Period 2) | 4.368 [4.310 to 4.425] | 4.442 [4.385 to 4.499]

4. Secondary Outcome: Knowledge of COVID-19 Prevention Message (Recall of ad, Intent to Travel, Mask Wearing and Beliefs About Travel)
Description: Facebook will ask a set of users in treated zip codes to answer four survey questions (each user answers only one question each). A small within-zip control group will be held from being treated, enabling comparisons between those who see the videos and those who don't. These questions will be asked a few days after the ad is shown on the User's feed and will include 1) recall of the ad; 2) intention of traveling over holiday; 3) intention of wearing a mask; and 4) beliefs about whether people should travel over holiday.
Time Frame: up to one month
Reporting Status: Not Posted

5. Secondary Outcome: Average Number of Tiles People Occupy (Mobility Measure)
Description: this measures each day "how much people move around by counting the number of level-16 Bing tiles they are seen in within a day. People seen in more tiles are probably moving around more, while people seen in fewer are probably moving around less. Each day take eligible people in a given region and compute the number of distinct tiles they were seen in." This is aggregated to the county level.
Time Frame: up to one month
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Eligible Participants Only Observed in a Single Level-16 Bing Tile (no Change in Movement)
Description: Facebook "Stay-put" data: this measures each day "the percentage of eligible people who are only observed in a single level-16 Bing tile (600m x 600m) during the course of a day" aggregated to they county level.
Time Frame: up to one month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed.
Arm/Group | High-Intensity Counties | Low-Intensity Counties
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/28/NCT04644328/Prot_SAP_000.pdf